CLINICAL TRIAL: NCT07379255
Title: Study Protocol for Evaluating the Efficacy of Postoperative Adjuvant Chemotherapy Drugs for Bladder Cancer Based on Organoid Technology.
Brief Title: Evaluation of Postoperative Adjuvant Chemotherapy Efficacy for Bladder Cancer Based on Organoid Technology.
Status: Recruiting | Type: Observational
Sponsor: Qilu Hospital of Shandong University (Other)
Collaborators: The Second Hospital of Shandong University (Other); Qianfoshan Hospital (Other); Shandong Provincial Hospital (Other Government); Shandong Province Third hospital (Other); Taian City Central Hospital (Other); Weifang People's Hospital (Other); Binzhou Medical University (Other); The Affiliated Hospital of Qingdao University (Other); Jining First People's Hospital (Other); Liaocheng People's Hospital (Other); Linyi People's Hospital (Other); Yantai Yuhuangding Hospital (Other); Zibo Central Hospital (Other Government); Dezhou Hospital Qilu Hospital of Shandong University (Other); Zaozhuang Municipal Hospital (Other); Qilu Hospital of Shandong University (Qingdao) (Other)
Responsible Party: Sponsor
Other Study IDs: KYLL-202411-008-2
Record Dates: First submitted 2026-01-23; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-12

CONDITIONS: Bladder Cancer
Keywords: Organoid; Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental group: Using tumor organoid drug sensitivity experiments to test the sensitivity of a patient's tumor cells to seven chemotherapy drugs and formulate a postoperative adjuvant chemotherapy plan.
  Interventions: Other: Organoid culture
- Control group: Select bladder cancer patients who underwent surgery during the same period and received postoperative adjuvant chemotherapy according to the empirical regimen as the control group.

INTERVENTIONS:
Other: Organoid culture — Organoid culture of tumor tissue obtained during patient surgery
  Groups: Experimental group

SUMMARY:
To evaluate the clinical efficacy of using tumor organoid drug sensitivity experiments to guide postoperative adjuvant chemotherapy in patients with muscle-invasive bladder cancer, and to assess the application value of tumor organoid drug sensitivity experiments in guiding individualized postoperative adjuvant chemotherapy for muscle-invasive bladder cancer.

DETAILED DESCRIPTION:
1. Research Background (Presenting the Rationale and Significance of This Study Based on Current Domestic and International Research)

   Bladder cancer is a malignant tumor originating from the bladder urothelium and ranks first in incidence among urogenital tumors in China. Among these, urothelial carcinoma is the most common, accounting for over 90% of bladder cancer cases [1]. Clinically, based on the depth of tumor invasion into the bladder wall and prognostic characteristics, bladder cancer is classified into non-muscle-invasive bladder cancer (NMIBC) and muscle-invasive bladder cancer (MIBC). MIBC constitutes approximately 20% of newly diagnosed bladder cancer cases [2-3], but its prognosis is significantly worse than that of NMIBC, with a 5-year overall survival (OS) rate of about 60%-70% [4-5].

   For patients with T2~T4a stage disease without distant metastasis, radical cystectomy (RC) is typically the standard treatment [2-3]. However, for high-risk patients with pT3-pT4 disease and/or pN+ M0 status, the 5-year survival rate following RC is only 25-35% [2, 6-8]. Therefore, combining systemic therapy with surgery plays a crucial role in reducing tumor progression rates. Multiple retrospective studies have shown that adjuvant chemotherapy after RC can delay recurrence and improve overall survival, providing clinical benefit. Skinner et al. [9] reported the first randomized trial, which demonstrated benefits for the adjuvant chemotherapy group in terms of disease-free survival (DFS) (51% vs. 34%) and overall survival (44% vs. 39%, n.s.) at 5 years. Another prospective randomized trial reported by Freiha et al. investigated the benefit of adjuvant CMV chemotherapy after RC in 50 patients with pT3b-T4, N0/+, M0 disease [10]. Consequently, guidelines recommend adjuvant chemotherapy for high-risk patients with pT3~pT4 disease or lymph node metastasis [11]. Currently, commonly used adjuvant chemotherapy drugs for bladder cancer include: cisplatin, gemcitabine, methotrexate, vinblastine, doxorubicin, paclitaxel... However, the variety of chemotherapy drugs and differing administration methods lead to treatment regimen selection often relying on physicians' clinical experience or specific research findings, lacking a unified standard, and being characterized by empiricism and randomness. Furthermore, some patients exhibit intrinsic resistance to certain chemotherapeutic agents. By the time clinical assessment confirms a patient's insensitivity to the applied drug, severe toxic side effects have often already occurred, potentially even leading to multi-drug resistance (MDR), thereby depriving the patient of the opportunity to choose alternative treatments. Therefore, how to evaluate chemotherapy response, avoid primarily resistant drugs, and directly select highly sensitive agents to achieve individualized chemotherapy has become a research hotspot.

   The realization of precise cancer treatment heavily relies on drug sensitivity testing. Through precise and individualized chemotherapy drug screening experiments, the most effective and least toxic treatment regimen can be identified for each patient before therapy begins. Developing patient-specific chemotherapy plans represents a new research direction for achieving precision treatment in bladder cancer and improving chemotherapy efficacy. Previously, the more commonly used preclinical models were traditional tumor cell lines and patient-derived xenograft (PDX) models. Tumor cell line culture is simple but insufficient to simulate the growth state of tumor cells within the patient's body, and drugs screened using this system have low clinical application value. Although PDX models can simulate in vivo tumor characteristics and preserve the tumor microenvironment, they have significant limitations, such as relatively low stable engraftment rates, long modeling and evaluation cycles (six months to one year), being time-consuming and labor-intensive, making them difficult to generate and utilize for high-throughput drug screening [12-15]. Therefore, to develop more personalized treatment and prevention strategies tailored to an individual's unique genetic, environmental, and lifestyle characteristics, minimizing risks and optimizing medical intervention outcomes, it is imperative to develop drug sensitivity testing models that can simulate the heterogeneity and complexity of bladder cancer.

   Organoids, specifically Patient-Derived Organoids (PDOs), are three-dimensional organotypic structures formed through the self-assembly of stem cells in vitro. They can differentiate into multiple organ-specific cell types and exhibit cell-cell interactions, cell-extracellular matrix interactions, and spatial organization, thereby recapitulating key functions and structures of real human organs in vitro while maintaining stable phenotypic and genetic characteristics. Compared to two-dimensional tumor cell lines and PDX models, tumor organoids can be cultured directly from a patient's own tissue. These organoids can effectively replicate key properties of the primary tumor, preserve the pathological morphology and biological mechanisms of the patient's tissue, retain tumor heterogeneity and a more authentic tumor microenvironment, and have the advantage of a short growth cycle [16]. This facilitates their use for sensitivity testing of chemotherapy drugs, molecularly targeted agents, anti-tumor antibodies, etc., in clinical cancer patients, predicting patient response to drugs, and holds potential for assisting clinical treatment decision-making.

   In 2018, a study published in Science reported the use of metastatic gastrointestinal cancer organoids for drug sensitivity testing [17]. This study compared and analyzed the differences in sensitivity to a series of targeted and chemotherapeutic drugs between 21 clinical patients and their corresponding PDOs, demonstrating strong consistency between the two. Compared with the patients' actual therapeutic outcomes, the PDO predictions were robust (sensitivity 100%, specificity 93%, positive predictive value 88%, and negative predictive value 100%). In 2020, Yao Y et al. [18] utilized biopsy tissues from 112 patients with locally advanced rectal cancer to construct 96 rectal cancer organoids. Eighty of these were selected to test their response to chemoradiotherapy, and the results showed that the sensitivity of rectal cancer organoids to chemoradiotherapy was highly consistent with the patients' clinical responses (sensitivity 78%, specificity 92%, accuracy 84%). Subsequently, consistency between PDO drug response and patient clinical response has also been observed in gastric cancer, breast cancer, and other tumors. Yan HHN et al. [19] established a gastric cancer organoid biobank using tumor tissues, adjacent normal tissues, and lymph node metastasis samples from 34 gastric cancer patients. Among them, two cases developed metastasis and received postoperative combination therapy with cisplatin and 5-FU, both showing good responses. Another case received preoperative chemotherapy and showed no response to postoperative capecitabine. Investigating the sensitivity of the PDOs from these three cases to the corresponding compounds revealed that the drug sensitivity of the PDOs was completely consistent with the clinical responses of the respective patients. Guillen KP et al. [20] generated PDX and PDO models from tumor samples of breast cancer patients with endocrine therapy resistance, recurrence, and metastasis, and performed histomorphological, genomic, and drug sensitivity analyses on these samples. The results indicated that both breast cancer PDX and PDO models highly recapitulated the tissue biology and genomics of their source tumors, and their responses to anti-tumor drugs were consistent. In this study, a patient with stage IIA triple-negative breast cancer developed liver metastasis approximately one year after undergoing preoperative chemotherapy and surgery. The researchers conducted in vitro and in vivo drug sensitivity tests on the constructed PDO and PDX models and found that the microtubule inhibitor eribulin had the best therapeutic effect. Based on this finding, the patient was guided to receive eribulin treatment, resulting in complete remission of the liver metastasis lasting nearly 5 months. These studies provide preliminary evidence for the potential of PDOs to guide clinical drug use for cancer patients. Additional research has shown that by comparing the drug response differences between normal organoids and PDOs, highly selective drugs can be identified, which may help reduce toxic side effects in clinical patients. Thus, conducting drug sensitivity testing via PDOs to discover the most suitable drug treatment plan will help improve clinical efficacy for cancer patients, reduce toxic side effects, the risk of drug resistance, and the likelihood of tumor recurrence, maximizing patient benefit.

   Therefore, leveraging patient-derived bladder cancer organoid models to conduct drug sensitivity testing for adjuvant chemotherapy in muscle-invasive bladder cancer, establishing a standardized bladder cancer organoid drug sensitivity testing system, and formulating screening criteria for bladder cancer organoid drug sensitivity testing, will enable the selection of optimal drug combination regimens. This approach can assist in developing novel individualized treatment plans for clinical application and undergo multi-center clinical validation, ultimately achieving true "avatar drug testing."
2. Research Question and Objectives (Elucidating the Scientific Questions and Research Objectives)

Research Question: This study employs a clinical controlled trial design to compare the one-year, three-year, and five-year overall survival rates between a patient group receiving interventions guided by organoid drug sensitivity testing and a patient group receiving traditional empirical treatment. Univariate Kaplan-Meier survival analysis will be used to compare the differences in recurrence rates between the two groups. The study aims to evaluate the application value of tumor organoid drug sensitivity experiments in guiding chemotherapy for bladder cancer.

Research Objective: By observing the clinical efficacy of adjuvant chemotherapy guided by the tumor organoid drug sensitivity method in bladder cancer patients, this study aims to evaluate the application value of tumor organoid drug sensitivity experiments in guiding individualized chemotherapy for bladder cancer.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age between 18 and 80 years, any gender; 2. For patients undergoing radical cystectomy, if the pathology meets inclusion criterion No. 3, tissue from the surgical specimen will be used for organoid culture; 3. Patients with pT3-pT4 and/or lymph node-positive MIBC who require adjuvant chemotherapy after surgery; 4. Patients who can tolerate platinum-based chemotherapy; 5. ECOG performance status of 0-2; 6. According to the investigator's judgment, able to comply with the study protocol, demonstrate good adherence, cooperate with the monitoring of adverse events and efficacy, and comply with follow-up; 7. Willing to voluntarily participate in this clinical trial, understand the study procedures, and have signed the informed consent form to participate in this study.

Exclusion Criteria:

* 1. Severe, life-threatening complications occurring after radical cystectomy, such as cardiovascular complications, renal failure, respiratory failure, liver failure, sepsis, pulmonary embolism, and major hemorrhage; 2. Individuals with immunodeficiency or impairment (e.g., patients with AIDS, or those receiving immunosuppressants or radiotherapy); 3. Participants known to be allergic to the study drug, similar drugs, or excipients, or those with an allergic constitution; 4. Individuals taking long-term corticosteroids or with a history of drug abuse or dependence; 5. Individuals planning pregnancy soon, currently pregnant, or breastfeeding; 6. Abnormal blood routine, liver and kidney function, and coagulation indices (considered abnormal if one or more of the following are met):

  1. Absolute neutrophil count (ANC) ≤ 1.5 × 10⁹/L;
  2. White blood cell count (WBC) ≤ 3.0 × 10⁹/L;
  3. Platelet count (PLT) ≤ 90 × 10⁹/L;
  4. Hemoglobin (HB) ≤ 90 g/L;
  5. Total bilirubin (TBIL) ≥ 1.5 × upper limit of normal (ULN) for the institution;
  6. Estimated glomerular filtration rate (eGFR) ≤ 30 ml/min/1.73m²;
  7. International normalized ratio (INR) and activated partial thromboplastin time (APTT) ≥ ULN (excluding patients on anticoagulant therapy, if considered clinically acceptable by the investigator); 7. Other factors that may cause the study to be prematurely terminated, such as:

  <!-- -->

  1. Patients with a past or current diagnosis of myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML);
  2. A history of clear neurological or psychiatric disorders, including epilepsy or dementia;
  3. Comorbidities that pose a serious risk to patient safety or could affect study completion (e.g., severe hypertension, diabetes, thyroid disorders, etc.);
  4. Other serious diseases requiring combined treatment or with severe laboratory abnormalities;
  5. Other serious diseases accompanied by familial or social factors that could affect participant safety, or the collection of data and samples;
  6. Uncontrolled comorbid conditions, including but not limited to ongoing or active infections requiring treatment, symptomatic congestive heart failure, unstable angina, or arrhythmias; 8. Individuals deemed by the investigator as unsuitable to participate in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who need to come to the research center for treatment of bladder cancer.
Sampling Method: Non-Probability Sample
Enrollment: 266 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
One-year OS ,Three-year OS and five-year OS | 2026.01.01-2030.12.31
  One-year overall survival rate, three-year overall survival rate, five-year overall survival rate.

SECONDARY OUTCOMES:
One-year PFS ,Three-year PFS and five-year PFS | 2026.01.01-2030.12.31
  One-year progression-free survival rate, three-year progression-free survival rate, five-year progression-free survival rate.

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Yes